CLINICAL TRIAL: NCT00327119
Title: A Phase 2 Multicenter Single Arm Clinical Trial of ABX EGF (Panitumumab) Monotherapy in Japanese Subjects With Metastatic Colorectal Cancer Who Developed Progressive Disease or Relapsed While on or After Prior Fluoropyrimidine, Irinotecan and Oxaliplatin Chemotherapy
Brief Title: Phase 2 Study of ABX-EGF (Panitumumab) in Japanese Subjects With M-colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20050216
Record Dates: First submitted 2006-05-16; First posted 2006-05-18 (Estimated); Last update posted 2009-09-14 (Estimated); Status verified 2009-09

CONDITIONS: Metastatic Colorectal Cancer
Keywords: EGFR; Fully human; Monoclonal antibody; Panitumumab; ABX-EGF; AMG954; Colorectal Cancer; Japan
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Panitumumab

INTERVENTIONS:
Drug: ABX-EGF (panitumumab)

SUMMARY:
The primary objective of this study is to assess the effect of treatment with ABX-EGF on best overall objective response rate by modified RECIST (confirmed complete or partial response) in Japanese subjects with metastatic colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic colorectal adenocarcinoma;
* Subjects must have become refractory to treatment or unable to continue treatment due to toxicity or other reasons during or after treatment with fluoropyrimidine, irinotecan and oxaliplatin for metastatic colorectal cancer including those who relapsed during or within 6 months from the completion of adjuvant therapy using the above agents; - Tumor expressing EGFr levels by immunohistochemistry (membrane staining must be positive in 1% of evaluated tumor cells).

Exclusion Criteria:

* Subjects who have prior experimental or approved antibodies (eg, bevacizumab) within 3 months before enrollment;
* Subjects who have prior EGFr targeting agents;
* Chemotherapy other than fluoropyrimidine (including oral agents such as UFT, TS-1), irinotecan, and oxaliplatin (or raltitrexed) for colorectal carcinoma in accordance with specified regimens (leucovorin and levamisole are not considered as chemotherapy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2006-04

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Muro K, Yoshino T, Doi T, Shirao K, Takiuchi H, Hamamoto Y, Watanabe H, Yang BB, Asahi D. A phase 2 clinical trial of panitumumab monotherapy in Japanese patients with metastatic colorectal cancer. Jpn J Clin Oncol. 2009 May;39(5):321-6. doi: 10.1093/jjco/hyp016. Epub 2009 Mar 14. PMID 19287023
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com